CLINICAL TRIAL: NCT00902122
Title: Open-Label, Multi-Center, Randomized, Active-Controlled, Phase 4 Study of rAd-p53 Gene Mono-Therapy, With Concurrent Radioactive Iodine , or Combination With Surgery in Subjects With Advanced Malignant Thyroid Tumors
Brief Title: rAd-p53 Gene Therapy for Advanced Malignant Thyroid Tumors
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen SiBiono GeneTech Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: rAd-p53-003
Record Dates: First submitted 2009-05-12; First posted 2009-05-14 (Estimated); Last update posted 2012-04-09 (Estimated); Status verified 2010-02

CONDITIONS: Advanced Malignant Thyroid Tumors
Keywords: p53 gene; thyroid; gene therapy; malignant tumors
MeSH Terms: conditions — Thyroid Diseases; Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): Five times of p53 gene intratumoral injection are given before surgery,then radical surgery will be conducted.
  Interventions: Drug: rAd-p53 gene
- 2 (Active Comparator): surgery
  Interventions: Procedure: surgery
- 3 (Experimental): p53 gene therapy
  Interventions: Drug: p53 gene therapy
- 4 (Active Comparator): p53 gene therapy plus radioactive iodine
  Interventions: Radiation: p53 gene therapy with radioactive iodine

INTERVENTIONS:
Drug: rAd-p53 gene — pre-surgery p53 gene treatment: 10exp12 virus particles per 3 days for 5 times
  Arms: 1
Procedure: surgery — removal of thyroid tumor
  Arms: 2
Drug: p53 gene therapy — p53 gene treatment: 10exp12 virus particles per 3 days for 10 times
  Arms: 3
Radiation: p53 gene therapy with radioactive iodine — p53 gene therapy with concurrent radioactive iodine pre-surgery p53 gene treatment: 10exp12 virus particles per 3 days for 10 times
  Arms: 4

SUMMARY:
This is multicenter, open-label, randomized, active-controled, phase IV study of local direct intra-tumor injection of rAd-p53 monotherapy, with concurrent radioactive iodine , or combination with surgery for treatment of advanced malignant thyroid tumors.

DETAILED DESCRIPTION:
Primary objectives of this study is to determine the efficacy profiles of rAd-p53 intra-tumor injection alone, with with concurrent radioactive iodine, or combination with surgery for treatment of advanced malignant thyroid tumors(stage III or IV) including target lesion complete response rate (LCR) and overall target lesion response rate (OLR), response duration (RD), and progress-free survival (PFS).

The secondary objectives of this study is to investigate overall response rate (OPCR) and overall complete response rate (OCR), overall survival (OS), ECOG, and safety of rAd-p53 monotherapy and combined with radioactive iodine,or surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Advanced stages of thyroid malignant tumors (stage III and VI)
2. At least one target tumor can be injected with study drug, the largest diameter greater than 2 cm
3. Histologically confirmed Oral and Maxillofacial malignant tumors
4. No prior chemotherapy, radiotherapy or biological tumor therapy in 2 weeks
5. Age: 18-85 years old
6. Expected to survive more 12 weeks
7. ECOG:0-2
8. Neutrophils≥1.5×109/L,Platelet≥ 80×109/L, Hb≥80g/L, bilitubin≤2mg/dl,ALT and AST ≤2×institutional upper limit of normal, Cr ≤1.5×institutional upper limit of normal,coagulation tests (PTT and INR) within normal range
9. Subject provided signed informed consent -

Exclusion Criteria:

1. Hypersensitive to study drug
2. Tumor(s) locate very close to important blood vessels and nerves, which affect injection
3. With a coagulation and bleeding disorder
4. With uncontrolled, intercurrent illness including but limited to symptomatic neurological illness, symptomatic congestive heart failure, unstable angina pectoris, significant pulmonary disease or hypoxia, or psychiatric illness
5. Local infection close to injection site or systemic infection
6. Pregnant or lactating
7. Principle investigator consider not suitable

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2009-05; Primary Completion 2012-08 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate | 3 years

SECONDARY OUTCOMES:
Progress-free survival | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jingqiang Zhu, MD,PhD, Principal Investigator — Department Of Thyroid and breast Surgery, West China hospital, Sichuan University
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China